CLINICAL TRIAL: NCT04746066
Title: Observational Study Multicentric Phamacological no Profit for the Treatment of Patients With Hemoglobinopathies and Rare Inherited Anemia Affected by Covid 19
Brief Title: Observational Study for Patients With Hemoglobinopathies and Rare Inherited Anemia and Covid 19
Status: Recruiting | Type: Observational
Sponsor: Società Italiana Talassemie ed Emoglobinopatie (Other)
Responsible Party: Sponsor
Other Study IDs: EMO AER COVID-19
Record Dates: First submitted 2021-02-02; First posted 2021-02-09 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Haemoglobinopathies
MeSH Terms: conditions — Hemoglobinopathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The COVID-19 pandemic is causing many deaths around the world, putting a strain on health services. Patients with pre-existing chronic conditions are most affected by the SARS-COV2 infection. Infectious complications are a common cause of mortality and one of the main causes of morbidity in all these diseases. The main objective of this project is the assessment of patients with thalassemia, drepanocytosis, other haemoglobinopathies and rares inherited anemias suffering from SARS-COV-2 to:

1. Obtain clinical and epidemiological data that can provide information on a possible increased vulnerability of these patients to SARS-COV-2 infection;
2. Sharing therapeutic approaches considering the lack of information about the treatment.

DETAILED DESCRIPTION:
The COVID-19 pandemic is causing many deaths around the world, putting a strain on health services. Patients with pre-existing chronic diseases are most affected by SARS-COV2 infection. Italy is one of the countries most involved. Thalassaemia, drepanocytosis, other hemoglobinopathies and inherited anemias are widespread in italy and the mediterranean area. Thalassaemia syndromes are characterized by different clinical forms with mutations in globin genes that cause the reduction or complete absence of synthesis of the globin chain. Transfusion therapy remains the basis of thalassaemia management. Based on the extent of the severity of anemia and clinical presentation, thalassaemia was classified as transfusion-dependent (TDT) and non-transfusion-dependent (NTDT). Transfusion inevitably contributes to iron overload, which is associated with secondary morbidity, including organ damage, especially heart, liver, bone tissue, and endocrine glands. In ntdt, comorbility is mainly related to chronic anemia and increased gastrointestinal iron adsorption.

Other inherited anaemias include a large group of pathologies such as: hyporegenerative anaemias, such as congenital diseritropoietic anaemia and diamond-blackfan anemia; anaemies from deficiency of red blood cell membrane proteins due to altered membrane structure, such as hereditary spherocytosis and hereditary ellipsocytosis, and impaired membrane transport function, such as hereditary stomatocytosis; anaemies due to enzymatic deficiency, the most frequent of which are pyruvate deficiency kinase and glucose-6 phosphate dehydrogenase; sideroblastic anaemias and all other hereditary microcytic anaemies such as irida. All these anemias are characterized by high phenotypic heterogeneity but in most cases chronic hemolytic anemia, iron overload and addiction transfusion are found (as a percentage of a variable of cases). Transfusion therapy remains the basis of the management of these anaemias along with splenectomy (not practicable in all these classes of anemia). As with thalassaemia syndromes, in such anaemias, we find secondary morbidity, such as heart, liver, and endocrine damage resulting from both chronic anemia and iron overload.

Infectious complications are a common cause of mortality and one of the main causes of morbidity in all these pathologies. The greater quantitative and functional quantities, the involve t and b lymphocytes, production of immunoglobulins, neutrophils and macrophages, chemotaxis and phagocytosis, as well as the complement system. Excess iron can alter the immune balance in favour of the growth of infectious organisms. Other factors include multiple transfusions, associated with constant allo-antigenic stimulation. A large percentage of adult patients are splenectomized and risk complications related to splenectomy such as capsuled bacterial infections and immune system changes; low levels of zinc, another immune regulator; iron chelation therapy, which predisposes to serious yersinia-like infections. The circulation of abnormal erythrocytes is the cause of another permanent immune stimulus. In addition, particularly in elderly patients, the coexistence of adrenal hypofunction makes the response to sepsis less effective.

However, we have no information on the vulnerability of patients with thalassaemia, drepanocytosis, other hemoglobinopathies and hereditary anemias to SARS-COV2 infection. In order to obtain more information useful to increase our knowledge, a retrospective survey has been planned.

The main objective of this project is the evaluation of patients with thalassaemia, drepanocytosis, other hereditary hemoglobinopathies and anaemias affected by SARS-COV2 to:

1. obtain clinical and epidemiological data that may dare information on a possible increased vulnerability of these patients to SARS-COV2;
2. share therapeutic approaches considering the lack of information about treatment.

This is an italian study of observational, pharmacological, non-interventional, retrospective, prospective and multicenter, non-profit cohort. Patients diagnosed with thalassaemia, drepanocytosis, other hemoglobinopathies and hereditary anaemia positive to the SARS-COV2 virus will be enlisted. Patient data from reference centers will be introduced into the card via a web service.

The scientific committee of the project has discussed and approved a set of data that will be collected by local centers and that will feed the data collection database.

The study will be launched in every Italian center that requires participation. The Italian Society of Thalassaemia and Hemoglobinopathies (SITE) in its role as a scientific reporting company for pathology and the Foranemia Foundation, a non-profit organization, makes available to the center of microcitemie, coordinator of the study, a special web space for online data collection assuming the costs.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients with an established diagnosis of thalassemia, sickle cell disease, other haemoglobinopathies and Rare Anemia inherit with a virological diagnosis of SARS-COV-2 infection.

EXCLUSION CRITERIA:

* nobody

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with an established diagnosis of thalassemia, sickle cell disease, other haemoglobinopathies and Rare Anemia inherit
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-03-31 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Covid 19 infection | through study completion, an average of 1 year
  Incidence of Covid 19 infections in patient with Hemoglobinopathies and Rare Anemia inherit

CONTACTS AND LOCATIONS:
Overall Officials: Gian Luca Forni, Principal Investigator — Ospedali Galliera - SSD Microcitemia, anemie congenite e dismetabolismo del ferro
Locations (2):
- Italy (2):
  - E.O. Ospedali Galliera, Genova
  - Ospedali Galliera - S.S.D. Microcitemia, anemie congenite e dismetabolismo del ferro, Genova

IPD SHARING:
Plan to Share IPD: Undecided